CLINICAL TRIAL: NCT07148024
Title: Effects of Endotracheal Tube Cuff Pressure Management on Upper Airway Edema During Cardiopulmonary Bypass in Coronary Artery Bypass Grafting: A Double-Blind, Randomized Controlled Trial
Brief Title: Cuff Pressure and Airway Edema in CABG With CPB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Engin Çetin (Other Government)
Responsible Party: Sponsor-Investigator, Engin Çetin, principal investigator, Kocaeli City Hospital
Organization: Kocaeli City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: KSH-ANREA-EC-03
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Airway Ultrasound; Airway Edema; Endotracheal Tube
Keywords: airway edema; coronary Bypass Greft Surgery; endotrecheal tube

STUDY DESIGN:
Intervention Model Description: Parallel assigment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ETT cuff pressure 0 mmHg (Active Comparator): ETT cuff pressure will be set to 0 mmHg
  Interventions: Device: ETT cuff pressure 0 mmHg
- ETT cuff pressure 20-30 mmHg (Active Comparator): ETT cuff pressure will be set to 20-30 mmHg
  Interventions: Device: ETT cuff pressure 20-30 mmHg

INTERVENTIONS:
Device: ETT cuff pressure 0 mmHg — In this group, the endotracheal tube (ETT) cuff pressure will be maintained at 0 mmHg during cardiopulmonary bypass (CPB)
  Arms: ETT cuff pressure 0 mmHg
Device: ETT cuff pressure 20-30 mmHg — In this group, the endotracheal tube (ETT) cuff pressure will be maintained at 20-30 mmHg during cardiopulmonary bypass (CPB)
  Arms: ETT cuff pressure 20-30 mmHg

SUMMARY:
This study investigates how endotracheal tube (ETT) cuff pressure management during cardiopulmonary bypass (CPB) in coronary artery bypass grafting (CABG) affects upper airway edema. Patients will be randomized into two groups: cuff pressure kept at 0 mmHg or maintained at 20-30 mmHg during CPB. Ultrasonography will be used to measure lateral pharyngeal wall thickness, tongue parameters, and other airway dimensions at predefined perioperative time points. The primary outcome is the change in lateral pharyngeal wall thickness as an indicator of airway edema. A total of 76 patients aged 18-80 years undergoing elective CABG with CPB will be enrolled. The results aim to clarify safe cuff pressure management strategies to reduce airway edema.

DETAILED DESCRIPTION:
Purpose This study aims to evaluate the effect of endotracheal tube (ETT) cuff pressure management during cardiopulmonary bypass (CPB) in coronary artery bypass grafting (CABG) surgery on the development of upper airway edema. Ultrasonography will be used to assess changes in lateral pharyngeal wall (LPW) thickness, tongue thickness, correlation between intravenous fluid volume at multiple perioperative time points.

Study Design

This is a prospective, randomized, double-blind, controlled clinical trial. Patients undergoing elective CABG with CPB will be randomly assigned into two groups:

Group 1: ETT cuff pressure maintained at 0 mmHg during CPB Group 2: ETT cuff pressure maintained at 20-30 mmHg during CPB Cuff pressures will be monitored with a manometer every 5 minutes and adjusted as needed. At the end of CPB, all patients will have standard cuff pressure (20-30 mmHg).

Outcomes Primary outcome: Changes in LPW thickness as a marker of upper airway edema assessed by ultrasonography at five time points (T0: Preoperative T1: Before initiation of CPB T2: At the end of CPB T3: 2nd postoperative hour).

Secondary outcomes: Changes in tongue thickness, correlation between intravenous fluid volume and airway edema.

Participation Approximately 76 patients (18-80 years, ASA III-IV) scheduled for elective CABG with CPB will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective coronary artery bypass grafting (CABG) surgery
* Aged 18-80 years
* ASA physical status class III-IV
* Providing written informed consent

Exclusion Criteria:

* History of difficult intubation
* Anatomical abnormalities of the upper airway
* Body mass index (BMI) > 35 kg/m²
* Acute respiratory tract infection
* Emergency surgeries

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Change in Lateral Pharyngeal Wall Thickness Measured by Airway Ultrasound | T0: Preoperative T1: Before initiation of CPB T2: At the end of CPB T3: 2nd postoperative hour
  To compare the effect of two different endotracheal tube (ETT) cuff pressures (0 mmHg vs. 20-30 mmHg) during cardiopulmonary bypass (CPB) in coronary artery bypass grafting (CABG) on upper airway edema. The degree of airway edema will be assessed by measuring changes in lateral pharyngeal wall thickness (in millimeters, mm) using ultrasound at predefined perioperative time points.

SECONDARY OUTCOMES:
ultrasonographic airway parameter -tongue width | T0: Preoperative T1: Before initiation of CPB T2: At the end of CPB T3: 2nd postoperative hour
  To compare the effects of two different endotracheal tube (ETT) cuff pressures (0 mmHg vs. 20-30 mmHg) during cardiopulmonary bypass (CPB) in coronary artery bypass grafting (CABG) on upper airway edema. The degree of edema will be assessed by changes in ultrasonographic airway parameter, specifically tongue width (mm), measured before and after the procedure
ultrasonographic airway parameter -tongue volume | T0: Preoperative T1: Before initiation of CPB T2: At the end of CPB T3: 2nd postoperative hour
  To compare the effects of two different endotracheal tube (ETT) cuff pressures (0 mmHg vs. 20-30 mmHg) during cardiopulmonary bypass (CPB) in coronary artery bypass grafting (CABG) on the development of upper airway edema, which will be assessed by ultrasonographic measurements of upper airway structures before and after the procedure, including tongue thickness (mm).Tongue thickness (millimeters, mm)
Correlation Between Intravenous Fluid Volume and Airway Edema | T0: Preoperative T1: Before initiation of CPB T2: At the end of CPB T3: 2nd postoperative hour
  To evaluate the correlation between the total intravenous fluid volume administered intraoperatively and the degree of airway edema, as measured by changes in ultrasonographic airway parameters (e.g., tongue thickness, pharyngeal wall thickness) at defined time points.

CONTACTS AND LOCATIONS:
Overall Officials: Engin Çetin, Principal Investigator — Kocaeli City Hospital
Locations (1):
- University of Health Sciences Kocaeli City Hospital, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aytac BG, Soyal OB. Ultrasonographic evaluation of the postoperative airway edema after robotic prostatectomy: a single center observational study. Eur Rev Med Pharmacol Sci. 2023 Sep;27(18):8505-8513. doi: 10.26355/eurrev_202309_33775. PMID 37782166